CLINICAL TRIAL: NCT01351753
Title: Does Reversal of Visceral Obesity by Drug Therapy Improve Vascular Function?
Brief Title: Drug Therapy Induced Weight Loss to Improve Blood Vessel Function in Subjects With Obesity
Acronym: REVIVE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Gary L. Pierce, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201012738
Record Dates: First submitted 2011-05-04; First posted 2011-05-11 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Obesity; Metabolic Syndrome X
Keywords: Obesity; Metabolic Syndrome X; Hypertension; Dyslipidemia; Impaired glucose tolerance
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Hypertension; Dyslipidemias; Glucose Intolerance | interventions — Metformin; Orlistat; Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Metformin (Active Comparator)
  Interventions: Drug: Metformin
- Metformin + Orlistat (Experimental)
  Interventions: Drug: Metformin; Drug: Orlistat
- Metformin + Topiramate (Experimental)
  Interventions: Drug: Metformin; Drug: Topiramate
- Topiramate (Experimental)
  Interventions: Drug: Topiramate
- Metformin + Topiramate + Orlistat (Experimental)
  Interventions: Drug: Metformin; Drug: Orlistat; Drug: Topiramate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin
  Arms: Metformin; Metformin + Orlistat; Metformin + Topiramate; Metformin + Topiramate + Orlistat
Drug: Orlistat
  Arms: Metformin + Orlistat; Metformin + Topiramate + Orlistat
Drug: Topiramate
  Arms: Metformin + Topiramate; Metformin + Topiramate + Orlistat; Topiramate
Drug: Placebo — Placebo pills and capsules for metformin, orlistat and topiramate
  Arms: Placebo

SUMMARY:
Obesity is common (>30% of US adults), contributes to substantial morbidity and mortality, but is difficult to treat. Partly this is due to the transient, arduous and modest nature of lifestyle interventions. Partly it is due to the limited efficacy and safety problems of existing pharmacotherapy. Only one drug, orlistat, is approved for long-term use in obesity; but its effects on weight are relatively small. There are drugs that have been approved for other diseases but which also reduce weight. One promising approach to treating obesity is combination therapy with orlistat and one or more of these other agents. The investigators propose an innovative approach to developing new therapies for obesity coupling the use of combination therapy with rigorous assessment of cardiovascular safety. Vascular function is a quantitative surrogate clinical endpoint that has been strongly and independently linked to future cardiovascular events.

Our hypothesis is that combination pharmacotherapy will reduce weight and improve vascular function in obese human subjects. The co-primary endpoints will be weight and vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 75 years
* Male or postmenopausal female
* BMI ≥ 30 kg/m2
* One or more major cardiovascular (CV) risk factors (hypertension, dyslipidemia, impaired glucose tolerance OR metabolic syndrome)

Exclusion Criteria:

* Congestive heart failure
* Renal impairment
* History of bariatric surgery (i.e. lap-band, Roux-en-Y or biliopancreatic diversion)
* Type I diabetes mellitus
* Weight loss > 10% in the past 6 months
* Recurrent nephrolithiasis
* Current treatment for seizure disorder
* Hepatic cirrhosis
* Current use of study medications
* Current use of oral estrogen
* History of smoking cessation in the past three months
* Current cholestasis or malabsorption syndrome
* Planned use of any herbal or over-the-counter supplements for weight loss
* History of allergic reactions to metformin, topiramate, orlistat or any of ingredients
* Medical conditions requiring continuous use of phosphodiesterase inhibitors and/or the inability to withhold phosphodiesterase inhibitors for 48 hours
* Participation in another clinical drug study within four weeks prior to this investigation.
* Participation in any other weight loss or rigorous exercise program.
* Any disease or condition that in the opinion of the investigator may interfere with completion of the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2014-01-09 (Actual); Study Completion 2014-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary L Pierce, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

REFERENCES:
- See also: Recruitment website — http://goo.gl/IHNtm

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Metformin only
- Metformin + Orlistat: Metformin
  Orlistat
- Metformin + Topiramate: Metformin
  Topiramate
- Topiramate: Topiramate only
- Metformin + Topiramate + Orlistat: Metformin
  Orlistat
  Topiramate
Period: Overall Study
Arm/Group | Metformin | Metformin + Orlistat | Metformin + Topiramate | Topiramate | Metformin + Topiramate + Orlistat | Placebo
Started | 22 | 20 | 21 | 21 | 21 | 23
Completed | 15 | 13 | 14 | 21 | 14 | 22
Not Completed | 7 | 7 | 7 | 0 | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Metformin + Orlistat | Metformin + Topiramate | Topiramate | Metformin + Topiramate + Orlistat | Placebo | Total
Number analyzed (Participants) | 22 | 20 | 21 | 21 | 21 | 23 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 21 | 21 | 19 | 23 | 125
  >=65 years | 1 | 0 | 0 | 0 | 2 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.04 (7.14) | 55.09 (7.46) | 54.19 (6.06) | 54.3 (9.05) | 56.14 (9.05) | 55.78 (7.89) | 55.13 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 14 | 13 | 13 | 16 | 83
  Male | 8 | 7 | 7 | 8 | 8 | 7 | 45
Region of Enrollment [Number; unit: participants]
  United States | 22 | 20 | 21 | 21 | 21 | 23 | 128
Weight [Count of Participants; unit: Participants] | 22 | 20 | 21 | 21 | 21 | 23 | 128

OUTCOME MEASURES:

1. Primary Outcome: Weight (% Change From Baseline)
Description: Weight obtained in the fasting state on a gowned subject.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: percentage of weight change
Groups:
- Metformin: Metformin
- Topiramate: Topiramate
Arm/Group | Metformin | Metformin + Orlistat | Metformin + Topiramate | Topiramate | Metformin + Topiramate + Orlistat | Placebo
Number analyzed (Participants) | 22 | 20 | 21 | 21 | 21 | 23
percentage of weight change | -10.9 [-14.4 to -7.2] | -10.5 [-14.0 to -6.9] | -14.0 [-17.3 to -10.5] | -12.2 [-15.6 to -8.6] | -16.7 [-20.3 to -13.0] | -6.7 [-10.5 to -2.7]

2. Secondary Outcome: Office Systolic Blood Pressure (mmHg Change From Baseline)
Description: Automated sphygmomanometry while sitting
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Metformin | Metformin + Orlistat | Metformin + Topiramate | Topiramate | Metformin + Topiramate + Orlistat | Placebo
Number analyzed (Participants) | 15 | 13 | 14 | 14 | 14 | 22
mmHg | -11.42 [-21.10 to -1.74] | -11.41 [-20.88 to -1.94] | -10.33 [-19.52 to -1.14] | -8.55 [-18.53 to 1.44] | -14.47 [-24.87 to -4.08] | -13.26 [-23.28 to -3.23]

3. Secondary Outcome: Waist (cm Change After 6 Months From Baseline)
Description: Body fat distribution measured using anthropometry (waist, neck and hip circumferences)
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: cm change
Arm/Group | Metformin | Metformin + Orlistat | Metformin + Topiramate | Topiramate | Metformin + Topiramate + Orlistat | Placebo
Number analyzed (Participants) | 15 | 13 | 14 | 14 | 14 | 22
cm change | -10.62 [-20.48 to -0.77] | -9.04 [-18.78 to -0.78] | -11.65 [-21.20 to -2.11] | -16.63 [-26.59 to -6.66] | -15.76 [-26.44 to -5.08] | -10.78 [-20.79 to -0.78]

4. Secondary Outcome: Carotid-femoral Pulse Wave Velocity (PWV)(Change After 6 Months From Baseline)
Description: Change in carotid-femoral pulse wave velocity (Sphygmocor).
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: meters/sec
Arm/Group | Metformin | Metformin + Orlistat | Metformin + Topiramate | Topiramate | Metformin + Topiramate + Orlistat | Placebo
Number analyzed (Participants) | 15 | 13 | 14 | 14 | 14 | 22
meters/sec | -1.09 [-2.96 to 0.78] | -1.56 [-3.47 to 0.36] | -1.29 [-3.13 to 0.55] | -0.24 [-2.13 to 1.64] | -0.46 [-2.48 to 1.56] | -0.74 [-2.98 to 1.50]

ADVERSE EVENTS:
Arm/Group | Metformin | Metformin + Orlistat | Metformin + Topiramate | Topiramate | Metformin + Topiramate + Orlistat | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20 | 0/21 | 0/21 | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/20 | 0/21 | 0/21 | 0/21 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No